CLINICAL TRIAL: NCT02323854
Title: The EMPrint™ Ablate and RESect Study in Patients With Metastatic Lung Tumors (EMPRESS)
Acronym: EMPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COVEMPR0437
Record Dates: First submitted 2014-12-13; First posted 2014-12-24 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer
Keywords: primary, recurrent, metastatic lung tumor, ablation
MeSH Terms: conditions — Lung Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ablation and Surgical Resection (Other): Ablation of lung tumor; followed by surgical resection of the ablation zone.
  Interventions: Device: Ablation; Procedure: Surgical Resection

INTERVENTIONS:
Device: Ablation — Percutaneous antenna will be placed into the target tumor under CT image guidance. Target tumor will be ablated and the antenna will be removed.
Procedure: Surgical Resection — The planned surgical resection of the lung tumor will be conducted as scheduled post ablation procedure.

SUMMARY:
Post market prospective, non-randomized, single-arm, multicenter study, designed to demonstrate dose response of an ablation system using a percutaneous approach in patients with primary, metastatic, or recurrent primary lung tumors.

DETAILED DESCRIPTION:
Primary Endpoint: Dose response as indicated by CT imaging, measurement of maximum diameter and volume.

Secondary Endpoint: Assessment of complete tumor ablation immediately post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject or authorized representative has provided informed consent.
* Subject is ≥18 years of age.
* At least one pulmonary metastasis ≤ 3.0 cm in maximum diameter resulting from distant primary cancers or at least one recurrence of primary lung cancer ≤ 3.0 cm in maximum diameter.
* Subject has been confirmed by a thoracic surgeon to be a surgical candidate for resection of the tumor targeted for ablation.
* Subject is willing and able to comply with all aspects of the treatment and evaluation schedule.
* ≥1 cm of tumor-free lung parenchyma between target tumor and pleura or fissure.

Exclusion Criteria:

* Pre-procedure Exclusion Criteria
* Contraindicated for surgery.
* Prolonged chest infection, defined as lung consolidation that requires hospitalization and greater than 10 days of antibiotics 30 days prior to surgery.
* Tumor abutting main stem bronchus, main pulmonary artery branches, esophagus and/or trachea.
* Tumor with pleural contact.
* Tumors located < 3 cm of staple lines or other metal objects.
* Patients diagnosed with GOLD Stage IV Emphysema.
* Uncontrollable coagulopathy
* Patients unable to tolerate discontinued use of anti-coagulants prior to and during the ablation procedure.
* Subject is pregnant (documented by a positive pregnancy test according to hospital standard practices) or is actively breast-feeding.
* Subject has participated in an investigational drug or device research study within 30 days of enrollment that would interfere with this study.
* The investigator determines that participation in the study may jeopardize the safety or welfare of the subject.
* Patients with implantable pacemakers and other electronic implants, in accordance with Instructions for Use (IFU).

Intraprocedural Exclusion Criteria

*Incidental intraprocedural finding that the subject no longer meets the study eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03-13 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damian E Dupuy, MD FACR, Principal Investigator — Lifespan-Rhode Island Hospital, Rhode Island, USA
Locations (4):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical College, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island
- University Hospital Frankfurt, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blackmon SH, Sterner RM, Eiken PW, Vogl TJ, Pua BB, Port JL, Dupuy DE, Callstrom MR. Technical and safety performance of CT-guided percutaneous microwave ablation for lung tumors: an ablate and resect study. J Thorac Dis. 2021 Dec;13(12):6827-6837. doi: 10.21037/jtd-21-594. PMID 35070367

RESULTS

PARTICIPANT FLOW:
Groups:
- Ablation and Surgical Resection: All subjects meeting the inclusion/exclusion criteria were enrolled into the study to receive microwave ablation from the Emprint™ Ablation System using a percutaneous approach in patients with metastatic or primary lung tumors.
  Percutaneous antenna will be placed into the target tumor under CT image guidance. Target tumor will be ablated and the antenna will be removed.
  Once the ablation procedure was completed, the scheduled surgical tumor resection was performed. Adverse event data was collected starting from the initial administration of anesthesia until conclusion of the first post-operative follow-up visit.
Period: Overall Study
Arm/Group | Ablation and Surgical Resection
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Ablation procedures were completed for 15 subjects, of which 15 (100%) completed the study. Primary and secondary endpoint results were available for 11 subjects.
Groups:
- Ablation and Surgical Resection: All subjects meeting the inclusion/exclusion criteria were enrolled into the study to receive microwave ablation from the Emprint™ Ablation System using a percutaneous approach in patients with metastatic or primary lung tumors.
  Percutaneous antenna will be placed into the target tumor under CT image guidance. Target tumor will be ablated and the antenna will be removed.
  Once the ablation procedure was completed, the scheduled surgical tumor resection was performed. Adverse event data were collected starting from the initial administration of anesthesia until conclusion of the first post-operative follow-up visit.
Arm/Group | Ablation and Surgical Resection
Number analyzed (Participants) | 15
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 58.9 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
  Germany | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Response
Description: Dose response was assessed by comparing actual ablation zone size and volume to predicted ablation zone size and volume prescribed by the physician using the Emprint™ Procedure Planning Application. Dose response was measured for each ablation zone using CT imaging immediately post ablation and prior to the surgical resection.
Time Frame: 1 Day
Population: Primary endpoint results were available for 11 subjects. Four out of 15 (26.6%) imaging sets were either not obtained or unable to be evaluated.
Measure: Mean (Standard Deviation); unit: percent difference
Arm/Group | Ablation and Surgical Resection
Number analyzed (Participants) | 11
percent difference
  % Change Ablation Zone Width (X) | -43.6 (18.8)
  % Change Ablation Zone Height (Y) | -15.1 (31.7)
  % Change Ablation Zone Depth (Z) | -32.8 (26.0)
  % Change (Actual Volume vs Predicted Volume) | -63.5 (26.3)
  % Change (Actual Calculated Vol. vs Predicted) | -57.7 (31.8)

2. Primary Outcome: Ablation Zone Shape
Description: Ablation width (X) / height (Y), ratio of 1 indicates spherical ablation zone shape
Time Frame: Same day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ablation and Surgical Resection
Number analyzed (Participants) | 11
Ratio | 0.6 (.2)

3. Secondary Outcome: Number of Participants With Complete or Incomplete Tumor Ablation
Description: The secondary endpoint was complete tumor ablation immediately post-procedure for each target tumor using histologic analysis. Complete ablation was defined as 100% nonviable tumor cells.
Time Frame: Same Day
Population: Secondary endpoint results were available for 11 subjects. For the secondary results, there were no tumors in four out of 15 samples (26.6%). Therefore, assessment of tumor cannot be made.
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation and Surgical Resection
Number analyzed (Participants) | 11
Participants
  Complete Ablation | 6
  Incomplete Ablation | 4
  Delayed Necrosis | 1

ADVERSE EVENTS:
Time Frame: 30 Days Post-procedure.
Arm/Group | Ablation and Surgical Resection
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation and Surgical Resection (N=15)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Guillain Barre Syndrome (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ablation and Surgical Resection (N=15)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
* Difficult to obtain the ablated tumor in resected sample
* Limitation to investigator to performing a single ablation
* Imaging was the only measure for dose response and was captured immediately post-procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT02323854/SAP_000.pdf
  • Study Protocol (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT02323854/Prot_001.pdf